CLINICAL TRIAL: NCT02858479
Title: Structural and Functional Brain Reorganization in Neuropathic Pain. Influences of the Loss of Sensitivity and the Atrophy Cortical on Activations Due to Stimulation Allodynic
Acronym: ALLO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: failure to recruit
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1308174; 2013-A01791-44 (Other: ANSM)
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with pain allodynic peripheral (Other)
  Interventions: Other: stimulation on painful area (area allodynic); Other: same stimulation on non-painful area; Radiation: MRI scan
- patients with pain allodynic central (Other)
  Interventions: Other: stimulation on painful area (area allodynic); Other: same stimulation on non-painful area; Radiation: MRI scan

INTERVENTIONS:
Other: stimulation on painful area (area allodynic) — these stimulations will be performed either with a brush, with a cold block or with forced air (cold air or air to ambient temp) : calibrated to induce pain bearable.
  stimulations for 6 seconds
Other: same stimulation on non-painful area — these stimulations will be performed either with a brush, with a cold block or with forced air (cold air or air to ambient temp) : calibrated to induce pain bearable.
  stimulations for 6 seconds
Radiation: MRI scan — 2 sessions for 10 minutes :
  * 11 controls stimulations for 6 s each spaced 20 s without stimulation.
  * 11 allodynic stimulations for 6 s each spaced 20 s without stimulation.

SUMMARY:
Neuropathic pain is a medical condition involving allodynia (painful perceptions in response to stimuli that normally are not) and spontaneous pain (occurring at rest, without stimulation).

This pain is secondary to nervous system injury affecting the sensory system. The lesion is either at the nerve endings of the spinal cord or brain. It induces a loss of sensitivity and reorganization of brain activity.

Previous studies in functional neuroimaging have focused on brain areas activated during allodynic stimuli compared to non-painful stimuli. The abnormalities have been reported, but it was not possible to conclude formally.

The objective of this study is to understand the brain dysfunction that induces allodynic pain considering the deafferentation of each patient and possible cortical losses.

ELIGIBILITY:
Inclusion Criteria:

* with neuropathic pain
* in the case of central lesions, the lesion must be unique and small
* treatment not stable opioid for one week
* consent signed

Exclusion Criteria:

* severe psychiatric history
* presence of an evolutive lesion, expansive, cancerous or tumorous underlying
* patient needing of opioid therapy
* contraindication at MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
the deafferentation rate | at baseline
  the deafferentation rate measured with thermo-test
gray matter rate | at baseline
  gray matter rate measured with MRI scan

SECONDARY OUTCOMES:
Analysis pain | at baseline
  Measured by visual analogue scale (0 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Roland PEYRON, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No